CLINICAL TRIAL: NCT05304910
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled, Single-dose Study Investigating the Safety, Tolerability and Pharmacokinetic Properties of Lu AG09222 in Healthy Caucasian, Chinese and Japanese Subjects
Brief Title: A Study Investigating the Movement of Lu AG09222 Into, Through, and Out of the Body of Healthy Caucasian, Chinese, and Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19825A
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lu AG09222 Low Dose (Experimental): Participants will receive a single dose of Lu AG09222 by subcutaneous (SC) injection on Day 1.
  Interventions: Drug: Lu AG09222
- Lu AG09222 High Dose (Experimental): Participants will receive a single dose of Lu AG09222 by SC injection on Day 1.
  Interventions: Drug: Lu AG09222
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo matching LU AG0922 by SC injection on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AG09222 — Lu AG09222 will be administered per schedule specified in the arm description.
  Arms: Lu AG09222 High Dose; Lu AG09222 Low Dose
Drug: Placebo — Placebo matching to Lu AG09222 will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The main goal of the study is to learn more about how the body absorbs and eliminates Lu AG09222 after a single dose is injected under the skin. Researchers will also investigate safety and tolerability effects of Lu AG09222 after administration.

ELIGIBILITY:
Inclusion Criteria:

* The participant is Japanese, defined as having 4 Japanese grandparents, or the participant is Caucasian, or the participant is Chinese, defined as having 4 Chinese grandparents.
* The participant has a body mass index (BMI) ≥18 and ≤28 kilograms (kg)/square meter (m^2) at the Screening Visit and at the Baseline Visit.

Exclusion Criteria:

* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.
* The participant has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin or adequately treated cervical intraepithelial neoplasia, that has not been in remission for >5 years prior to the first dose of investigational medicinal product (IMP).
* The participant has had major surgery (excluding laparoscopic cholecystectomy or uncomplicated appendectomy) <6 months prior to the first dose of IMP.
* The participant has previously been dosed with Lu AG09222.
* The participant has a history of severe drug allergy or hypersensitivity.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Area Under the Lu AG09222 Serum Concentration-Time Curve (AUC) From Zero to Infinity (AUC0-inf) | Day 1 (predose) to Day 84
Maximum Observed Concentration (Cmax) of Lu AG09222 | Day 1 (predose) to Day 84
Apparent Elimination Half-Life (t½) of Lu AG09222 | Day 1 (predose) to Day 84
Time to Maximum Observed Concentration (tmax) | Day 1 (predose) to Day 84
Apparent Total Clearance (CL/F) | Day 1 (predose) to Day 84
Apparent Volume of Distribution (Vz/F) | Day 1 (predose) to Day 84

SECONDARY OUTCOMES:
Number of Participants With Specific Anti-Lu AG09222 Antibodies (Anti-Drug Antibodies [ADA]) | Day 1 (predose) to Day 84
Number of Participants With Specific ADA-Positive Samples for Neutralizing Antibodies (NAb) | Day 1 (predose) to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- PAREXEL International, Glendale, California, United States